CLINICAL TRIAL: NCT01031290
Title: Pilot Study Repetitive Transcranial Magnetic Stimulation (rTMS) in Cannabis Craving
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Maryland (Other)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999909443; 09-DA-N443
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-02-27

CONDITIONS: Cannabis Use
Keywords: Cue-Induced Craving; Cannabis; Functional Magnetic Resonance Imaging (fMRI); Repetitive TMS (rTMS); Cannabis Craving
MeSH Terms: conditions — Marijuana Abuse | interventions — Transcranial Magnetic Stimulation

ARMS (2):
- Group A (Experimental): Active TMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Group B (Sham Comparator): Sham TMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — daily sessions for 5 days

SUMMARY:
Background:

* Cannabis, also known as marijuana, is a commonly abused drug. There is no approved medication to treat cannabis addiction. The desire to use cannabis often increases when seeing others use it or seeing pictures of it. Researchers are interested in determining which parts of the brain are active when looking at pictures associated with cannabis.
* Repetitive transcranial magnetic stimulation (rTMS) uses magnetic pulses to stimulate the brain. These pulses can change activity in parts of the brain. Researchers are interested in determining whether rTMS can decrease activity in the parts of the brain that respond to cannabis, and thereby lessen cravings for cannabis.

Objectives:

- To determine whether transcranial magnetic stimulation can lower craving for cannabis when people who use cannabis are shown images that increase craving.

Eligibility:

- Individuals 18 years of age and older who are physically healthy and currently use cannabis (at least 3 times weekly for the past 2 years).

Design:

* The study will involve eight visits over 3 weeks, with each visit lasting 1 to 2 hours.
* Participants will have an initial assessment about cannabis use and provide blood and urine samples before beginning the study.
* Participants will have three magnetic resonance imaging (MRI) brain scans. The first MRI scan will look at the structure of the brain at rest. During the other two scans, participants will look at images related to and not related to cannabis use.
* The rTMS sessions (with either actual TMS or inactive [sham] TMS) will be held daily for 5 consecutive days. During these testing visits, researchers will ask questions related to drug use and craving, and collect urine and breath samples for further study.
* Participants will have two follow-up visits, 1 week and 2 weeks after the rTMS sessions, to evaluate memory and mood, and one final MRI brain scan at the end of the study.

DETAILED DESCRIPTION:
Primary objective:

Repetitive transcranial magnetic stimulation (rTMS) provides a non-invasive means of altering brain neural activity. This pilot study will test whether 5 days of rTMS reduces cue-induced cannabis craving and use in cannabis users.

Hypothesis:

We predict that active rTMS will significantly lower craving for cannabis compared with sham rTMS.

Study population:

Thirty healthy adult cannabis users (for at least 2 years, currently averaging 3 times weekly) with no other major psychiatric disorders except nicotine dependence (DSM IV criteria) will be recruited from the community.

Design:

Following a baseline phase to evaluate subject characteristics, subjects will be randomly assigned to receive 5 days of active or sham rTMS. rTMS at 1 Hz and strength 120% of the motor threshold will be applied to the dorsolateral prefrontal cortex (DLPFC) using a figure 8 coil , beginning 1 second after presentation of a cannabis-associated visual cue and lasting for 30 seconds. Brain site localization will use a computerized navigation system based on structural MRI scans obtained before the first session. Each rTMS session (lasting around 31 minutes) will consist of 54 trials (cue presentations): 36 with cannabis-associated cues and 9 each with non-drug-associated positive or neutral cues. No rTMS will be administered with the non-cannabis-associated cues. Subjects return for follow-up assessments one and two weeks after the final rTMS session.

Outcome measures:

The primary outcome measure will be cannabis craving assessed by the Marijuana Craving Questionnaire and visual analog scales before and after every rTMS session and at one- and two-week follow-up. Secondary outcome measures will be self-reported cannabis use and urine drug testing at each rTMS session and follow-up visit, and changes in regional brain responses to cannabis-associated visual cues assessed by fMRI done before and after the 5 rTMS sessions.

Benefits:

The future benefit to society may be development of better methods for treatment of cannabis addiction.

Risks:

The primary risks from rTMS are transient headache, scalp discomfort, decreased spatial recognition memory, and hearing loss (minimized by wearing ear plugs). Seizures are very rare when rTMS is administered within accepted safety guidelines and individuals at increased risk of seizures are excluded. The risk of inducing a manic episode is minimized by excluding individuals with a history of non-drug-induced mania/hypomania.

ELIGIBILITY:
-INCLUSION CRITERIA:

i) Eighteen to sixty-five years of age

ii) Cannabis user for at least 2 years, currently averaging 3 times weekly

iii) Reading level of at least 6th grade, based on the Wide Range Achievement Test (WRAT)

iv) Ability to give valid informed consent

v) Right-handed

vi) If the subject is female, of childbearing potential, and sexually active, she agrees to use a medically acceptable form of contraception, and not become pregnant for the duration of the study. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. Female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use either: (1) contraceptive pill or IUD or depot hormonal preparation (ring, injection, implant); and/or (2) a barrier method of contraception such as diaphragm, sponge with spermicide, or condom. Women who are not sexually active do not have to agree to use one of the acceptable contraception methods. Contraceptive measures will be reviewed with female subjects at each visit prior to the rTMS treatment

vii) Self-report experiencing cannabis craving when exposed to cannabis-associated cues

EXCLUSION CRITERIA:

i) Personal or first-degree family history of any clinically defined neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness.

ii) Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head that cannot be safely removed.

iii) Metal shrapnel or bullet in the head or body including metal shavings.

iv) Current use of any investigational drug or of any medications with anti or pro-convulsive action

v) Increased intracranial pressure (lowers seizure threshold)

vi) Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania

vii) History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.

viii) Pregnant or nursing women or women with reproductive potential not using an acceptable form of contraception.

ix) Any history of seizure

x) Current dependence (DSM-IV criteria) on substances other than cannabis or nicotine.

xi) Claustrophobia making them unable to tolerate lying in the MRI scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08-19; Primary Completion 2012-01-31 (Actual); Study Completion 2012-02-27 (Actual)

PRIMARY OUTCOMES:
Cannabis craving by Marijuana Craving Questionnaire and visual-analogue scales. | 2 weeks

SECONDARY OUTCOMES:
Cannabis use by urine drug testing and self-report; Safety and tolerability, using side-effects checklist. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Allen EA, Pasley BN, Duong T, Freeman RD. Transcranial magnetic stimulation elicits coupled neural and hemodynamic consequences. Science. 2007 Sep 28;317(5846):1918-21. doi: 10.1126/science.1146426. PMID 17901333
- [Background] Bestmann S, Baudewig J, Siebner HR, Rothwell JC, Frahm J. Functional MRI of the immediate impact of transcranial magnetic stimulation on cortical and subcortical motor circuits. Eur J Neurosci. 2004 Apr;19(7):1950-62. doi: 10.1111/j.1460-9568.2004.03277.x. PMID 15078569
- [Background] Brody AL, Mandelkern MA, London ED, Childress AR, Lee GS, Bota RG, Ho ML, Saxena S, Baxter LR Jr, Madsen D, Jarvik ME. Brain metabolic changes during cigarette craving. Arch Gen Psychiatry. 2002 Dec;59(12):1162-72. doi: 10.1001/archpsyc.59.12.1162. PMID 12470133